CLINICAL TRIAL: NCT03275948
Title: Effects of Whole Grain on Cognitive Performance and Mood, and the Relationships to Cardiometabolic Risk Markers
Brief Title: Effects of Whole Grain Rye on Metabolic Risk Markers and Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Anne Nilsson, Associate professor, PhD, Lund University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2016/487
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Metabolic Disorders and Cognitive Decline
MeSH Terms: conditions — Metabolic Diseases; Cognitive Dysfunction | interventions — Whole Grains

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whole grain (Experimental)
  Interventions: Other: whole grain
- refrence (Other): white wheat based product
  Interventions: Other: reference

INTERVENTIONS:
Other: whole grain — whole grain rye
  Arms: whole grain
Other: reference — white wheat bread
  Arms: refrence

SUMMARY:
The purpose of the study is to investigate, in healthy middle age subjects, effects of whole grain rye on cognitive functions, mood, and cardiovasculair risk markers

ELIGIBILITY:
Inclusion Criteria:

* healthy
* BMI 19-28
* plasma glucose < 6.1 mmol/L
* non smooker

Exclusion Criteria:

* known metabolic diseases
* known gastrointestinal disorders
* known cognitive decline.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
cognitive performance | postprandial 0-180 min after breakfast
  test of working memory capacity

SECONDARY OUTCOMES:
glucose tolerance | 0-180 min after breakfast
  postprandial glucose concentrations

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sandberg JC, Bjorck IME, Nilsson AC. Impact of rye-based evening meals on cognitive functions, mood and cardiometabolic risk factors: a randomized controlled study in healthy middle-aged subjects. Nutr J. 2018 Nov 6;17(1):102. doi: 10.1186/s12937-018-0412-4. PMID 30400947